CLINICAL TRIAL: NCT02437838
Title: Optimizing Drug Doses to Improve Outcomes of Critically Ill Patients
Brief Title: Optimizing Drug Doses in Critically Ill
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0455
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Traumatic Brain Injury; Kidney Functional
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The primary objectives of this study are to examine whether augmented renal clearance (ARC) compromises renally eliminated drug therapeutic serum concentrations in patients with traumatic brain injury (TBI) and to estimate the optimal dose needed to achieve therapeutic serum concentrations of the probe medication levetiracetam in patients with TBI.

DETAILED DESCRIPTION:
Purpose: The primary objectives of this study are to examine whether augmented renal clearance compromises renally eliminated drug therapeutic serum concentrations in patients with traumatic brain injury (TBI) and to estimate the optimal dose needed to achieve therapeutic serum concentrations of the probe medication levetiracetam in patients with TBI.

Participants: The population will be comprised of patients with traumatic brain injury requiring levetiracetam for seizure prophylaxis admitted to the neurosciences intensive care unit

Procedures (methods): This is a multi-center, prospective, non-randomized pharmacokinetic study in patients with TBI. In patients who meet the inclusion criteria, a 12-hour urine collection for measuring creatinine clearance levetiracetam urine concentrations will be performed daily for 7 days. Serum levetiracetam concentrations will be obtained twice daily for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years
2. Patients with TBI requiring levetiracetam for seizure prophylaxis
3. Anticipated length of stay in the SICU or NSICU > 48 hours
4. Informed consent provided by the patient's designated medical proxy

Exclusion Criteria:

1. Pregnancy
2. Patients with renal dysfunction (CKD stages 3 - 5 and/or SCr > 1.4 mg/dL)
3. Patients receiving renal replacement therapy
4. Brain death or suspected imminent brain death within the next 48 hours
5. Patients with history of nephrectomy or renal transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients with traumatic brain injury requiring levetiracetam admitted to the University of North Carolina Intensive Care Unit and University of Kentucky Chandler Medical Center Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To examine whether ARC compromises renally eliminated drug therapeutic serum concentrations in patients with TBI (urine collections/ two levetiracetam serum concentrations, to measure creatinine clearance and therapeutic drug concentrations) | Daily 12-hour urine collections and two levetiracetam serum concentrations will be performed to directly measure creatinine clearance and therapeutic drug concentrations up to day 7 of ICU stay

SECONDARY OUTCOMES:
To estimate the optimal dose needed to achieve therapeutic serum concentrations of the probe medication levetiracetam in patients with TBI | Data will be obtained during study period of up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Morbitzer, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Cook AM, Hall K, Kolpek JH, Morbitzer KA, Jordan JD, Rhoney DH. Enhanced renal clearance impacts levetiracetam concentrations in patients with traumatic brain injury with and without augmented renal clearance. BMC Neurol. 2024 Jan 2;24(1):12. doi: 10.1186/s12883-023-03515-w. PMID 38166710